CLINICAL TRIAL: NCT05635591
Title: KSD-101 Therapy for EBV-associated Haematologic Neoplasms: an Exploratory Clinical Trial
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tongji Hospital (Other)
Collaborators: Kousai Bio Co., Ltd. (Other)
Responsible Party: Principal Investigator, Chunrui Li, Principal Investigator, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSD-101-CR001
Record Dates: First submitted 2022-11-14; First posted 2022-12-02 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: EBV-associated Haematologic Neoplasms
Keywords: EBV; haematologic neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KSD-101 (Experimental)
  Interventions: Biological: Autologous monocyte - derived DCs pulsed with EBV antigen

INTERVENTIONS:
Biological: Autologous monocyte - derived DCs pulsed with EBV antigen — Patients will receive approximately （5-10）x10^6 DC vaccine via subcutaneous injections bi-weekly,totally 3-5 times.

SUMMARY:
The primary objectives of this study is to evaluate the tolerability and safety of KSD-101 in Patients with EBV-associated haematologic neoplasms, observe the dose-limiting toxicity (DLT) and and to explore the maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his legal guardian participated voluntarily and signed the informed consent form.
2. A patient aged 18 - 70 years ( inclusive ) on the day of signing the informed consent form, male or female.
3. A patient who is diagnosed with EBV - associated haematologic neoplasms，and fail to respond or relapse after conventional treatment, or voluntarily choose therapeutic DC vaccines as the salvage therapy.
4. ECOG performance score 0 - 1.
5. Meet apheresis or intravenous blood collection criteria and no other contraindications.
6. Adequate organ function:Hematology: neutrophils of ≥1×10^9 /L , hemoglobin of ≥ 70 g / L, platelets of ≥ 50 ×10^9 / L. Liver function: ALT, AST ≤ 3 × ULN and TBIL ≤ 1.5 × ULN.Renal function: creatinine ≤ 1.5 × ULN. Cardiac function: left ventricular ejection fraction LVEF ) ≥ 40%. Coagulation function: fibrinogen ≥ 1.0 g / L, activated partial thromboplastin time ( APTT ) ≤ 1.5 × ULN, prothrombin time ( PT ) ≤ 1.5 × ULN.
7. A patient who has a lymph node area where subcutaneous injection can be performed.

Exclusion Criteria:

1. A patient who has received any anticancer therapy such as chemotherapy, radiotherapy or immunotherapy (eg, immunosuppressive drugs) within one month prior to screening.
2. A female patient who is pregnant (positive urine/blood pregnancy test) or breastfeeding, or a male/female patient who plans to conceive in recent 1 year.
3. A patient who has positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), with positive titer of hepatitis B virus (HBV) DNA in peripheral blood; or has positive hepatitis C virus (HCV) antibody, hepatitis C virus (HCV) RNA in peripheral blood, human immunodeficiency virus (HIV) antibody, or syphilis.
4. A patient who has central nervous system disorders (e.g., brain oedema, hormonal intervention indicated, or progression of brain metastases).
5. Patients had an uncontrollable infectious disease within the first 4 weeks of enrollment（ except the CTCAE toxicity grade is less than 2 of genitourinary infections and upper respiratory tract infections , EBV infection）
6. A patient who has serious underlying diseases (such as cardiovascular disease, respiratory disorder, renal insufficiency, coagulation disorder, autoimmune disease or immunodeficiency disease, etc.).
7. A patient who has had other active malignancies within the last 3 years, unless curable and clearly cured, such as basal or squamous cell carcinoma, carcinoma in situ of cervix or breast, etc.
8. A patient who has received prophylactic live or live-attenuated vaccines within 4 weeks prior to screening
9. A patient who has participated in other clinical studies within 4 weeks prior to screening
10. A patient who has a prior history of serious drug allergy or penicillin allergy.
11. A patient who has a history of drug abuse/addiction.
12. A patient who has any conditions resulting in ineligibility for enrollment as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) by dose group | 1 years after DC Vaccines injection
  Dose limiting toxicity will be assessed after injection in each dose group
Incidence of maximally tolerated dose (MTD) by dose grouphaematologic neoplasms | 1 years after DC Vaccines injection
  Maximally tolerated dose will be assessed after injection in each dose group
Type and incidence of adverse events (AEs) and serious adverse events (SAEs) by dose group | 1 years after DC Vaccines injection
  Calculate type and incidence of adverse events (AE), serious adverse event (SAE), including those happened after injection, those related to study drug, or those that led to withdrawal from the study. They will also be aggregated by systematic organ classification (SOC), preferred term (PT), and severity.

SECONDARY OUTCOMES:
EBV-DNA load | 1 years after DC Vaccines injection
  The load levels of EBV-DNA will be detected at each time point
Objective response rate (ORR) | 1 years after DC Vaccines injection
  The percentage of participants who achieved PR or better response
Disease control rate (DCR) | 1 years after DC Vaccines injection
  The percentage of participants who achieved SD or better response
Duration of response (DOR) | 1 years after DC Vaccines injection
  DOR will be calculated among responders (with a PR or better response) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease
Progression-free survival (PFS) | 1 years after DC Vaccines injection
  The time from the start of CAR-GPRC5D treatment for the participants to the first time of disease progression or death for any reason
Overall survival (OS) | 1 years after DC Vaccines injection
  OS is measured from the date of the initial injection of DC Vaccines to the date of the participant's death
Levels of EBV-specific CD8+ T cells | 1 years after DC Vaccines injection
  EBV-specific CD8+ T cells in peripheral blood will be assessed to monitor changes
Levels of B cells | 1 years after DC Vaccines injection
  B cells in peripheral blood will be assessed to monitor changes
Levels of NK cells | 1 years after DC Vaccines injection
  NK cells in peripheral blood will be assessed to monitor changes

CONTACTS AND LOCATIONS:
Overall Officials: Li Chunrui, Principal Investigator — Tongji Hospital
Locations (1):
- Li Chunrui, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided